CLINICAL TRIAL: NCT00184652
Title: The Effect of Norditropin® on Nutritional Status in Adult Patients in Chronic Haemodialysis
Brief Title: Growth Hormone Treatment in Adult Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1606-1442
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Asia, Europe, and Middle East. Adult patients with chronic kidney disease are treated with growth hormone to assess effect on nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients

Exclusion Criteria:

* Diabetes Mellitus
* Severe and Malignant diseases
* Patients in Intensive Care Units

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change in surrogate markers of nutrition | After 6 months treatment

SECONDARY OUTCOMES:
Quality of Life
Other markers of nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR 1452), Study Director — Novo Nordisk A/S
Locations (26):
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus N
  - Novo Nordisk Investigational Site, København Ø
  - Novo Nordisk Investigational Site, Odense
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Heidelberg
- Novo Nordisk Investigational Site, Hong Kong, Hong Kong
- Israel (6):
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Ramat Gan
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tzriffin
- Poland (3):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Wołomin
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Gothenburg, Sweden
- Novo Nordisk Investigational Site, Bern, Switzerland
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Feldt-Rasmussen B, Lange M, Sulowicz W, Gafter U, Lai KN, Wiedemann J, Christiansen JS, El Nahas M; APCD Study Group. Growth hormone treatment during hemodialysis in a randomized trial improves nutrition, quality of life, and cardiovascular risk. J Am Soc Nephrol. 2007 Jul;18(7):2161-71. doi: 10.1681/ASN.2006111207. Epub 2007 Jun 6. PMID 17554147
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com